CLINICAL TRIAL: NCT01170026
Title: Individual and Family Motivational Interviews for Substance Using Truant Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1 R34 DA0029871
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Substance Use
Keywords: substance use; adolescents; intervention; truancy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Check-up/Individual MI (Experimental): Two session motivational intervention to improve parent monitoring and communication with respect to adolescent risk behavior especially substance use plus 2 session Individual Motivational Intervention for the adolescent
  Interventions: Behavioral: Family Check-up/ Individual MI
- Psychoeducation (Active Comparator): Two sessions of psychoeducation for parents regarding adolescent risk behaviors especially substance use
  Interventions: Behavioral: Individual and family psychoeducation

INTERVENTIONS:
Behavioral: Family Check-up/ Individual MI — The 2-session intervention protocol consists of an individual motivational interview plus the Family Check-Up (Dishion & Kavanagh, 2003), a family based motivational interview. The experimental protocol provides a thorough assessment of both individual and family strengths and weaknesses with respect to substance use prevention and school attendance/performance.
  Other Names: (Family Check-up)
  Arms: Family Check-up/Individual MI
Behavioral: Individual and family psychoeducation — Families in PE will return for the same number of visits as the IMI and FCU sessions of the IMI/FCU condition. An interventionist will review a set of educational materials with the parents regarding teen SU use, truancy and risk behaviors and parenting a teenager. A similar set of materials will be reviewed with the adolescent
  Other Names: (Psychoed)
  Arms: Psychoeducation

SUMMARY:
This application will provide a test of one potential model for adding substance use assessment and brief intervention into a truancy court program. The primary goal of this study is to determine whether a motivational intervention will reduce substance use among adolescents referred to truancy court for school attendance problems. In this treatment development application, an open trial with 20 families referred by truancy court will first be conducted. This trial will be used to adapt an existing motivational intervention to include material relevant to school attendance and performance. Then 100 families participating in the Rhode Island Truancy Court Program with adolescents between the ages of 13-16 years who report using substances will be randomly assigned to receive the experimental intervention plus standard truancy court procedures or psychoeducation plus standard truancy court procedures. The 2-session intervention protocol consists of an individual motivational interview plus the Family Check-Up (Dishion & Kavanagh, 2003), a family based motivational interview. The experimental protocol provides a thorough assessment of both individual and family strengths and weaknesses with respect to substance use prevention and school attendance/performance. Follow-up interviews will be conducted at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 13-16 at the start of the project and living at home with at least one parent/guardian,
2. t- score of 70 or above on one of the diagnostic-oriented scales (internalizing or externalizing problems) on the Child Behavior Checklist (i.e. reach the clinical cut-off),
3. the child must report 6 or more incidences of substance use in the last 90 days,
4. parental consent and child assent are obtained.

Exclusion Criteria:

1. adolescent meets diagnostic criteria for substance dependence suggesting need for more intensive services,
2. the family is not able to speak and understand English or Spanish well enough to complete study procedures.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown Medicl School
Locations (1):
- Brown University, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Family Court
Period: Overall Study
Arm/Group | Family Check-up/Individual MI | Psychoeducation
Started (Completed 6 months) | 34 (Followed up for 6 months) | 35 (Followed up for 6 months)
Completed | 30 (Completed 6 months) | 33 (Completed at 6 months)
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat analyses were used
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Check-up/Individual MI | Psychoeducation | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.4) | 16.0 (1.2) | 15.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 21 | 27 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 23 | 18 | 41
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Use Days in Past 90 Days
Description: Number of Days in which a Participant Responded "Yes" to Marijuana use in the Past 90 Days" range = 0 to 90; higher scores indicate more marijuana use
Time Frame: 3 Month Follow-Up and 6 month follow-up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Family Check-up/Individual MI | Psychoeducation
Number analyzed (Participants) | 34 | 35
days
  Baseline | 35 (29) | 45 (39)
  3-month follow-up | 27 (35) | 41 (36)
  6-month follow-up | 21 (28) | 41 (35)

2. Primary Outcome: Alcohol Use Days in Past 90 Days
Description: If a Participant Responded "Yes" to Alcohol use in the Past 90 Days" ; yes /no
Time Frame: 3 and 6 Month Follow-Up
Measure: Count of Participants; unit: Participants
Arm/Group | Family Check-up/Individual MI | Psychoeducation
Number analyzed (Participants) | 34 | 35
Participants
  Baseline | 20 | 26
  3-month follow-up | 8 | 17
  6-month follow-up | 11 | 18

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Family Check-up/Individual MI | Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

LIMITATIONS AND CAVEATS:
The small sample size suggests that the findings may not be stable. Substance use was self-reported and not corroborated by secondary observers, with the exception of the UDS data at 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT01170026/Prot_SAP_000.pdf